CLINICAL TRIAL: NCT01047787
Title: Breathing Disorders in Patients With Congestive Heart Failure: Gender and Mortality Impact
Brief Title: Breathing Disorders in Patients With Congestive Heart Failure
Status: Completed | Type: Observational
Sponsor: University of Sao Paulo (Other)
Responsible Party: University of Sao Paulo, Rogerio Santos da Silva
Other Study IDs: 823/01
Record Dates: First submitted 2007-05-15; First posted 2010-01-13 (Estimated); Last update posted 2010-01-13 (Estimated); Status verified 2007-05

CONDITIONS: Congestive Heart Failure
Keywords: Sleep apnea; Cheyne-Stokes Respiration; Congestive Heart Failure
MeSH Terms: conditions — Heart Failure; Sleep Apnea Syndromes; Cheyne-Stokes Respiration

STUDY DESIGN:
Observational Model: Case-Crossover | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (1):
- CHF Patients: Congestive Heart Failure Patients
  Interventions: Other: Polysomnography

INTERVENTIONS:
Other: Polysomnography — examination for sleep disorders

SUMMARY:
The investigators prospectively evaluated 89 consecutive outpatients (29 female) with stable congestive heart failure. The presence of sleep disordered breathing (SDB) and Cheyne-Stokes respiration (CSR) while awake were investigated by overnight polysomnography. Males and females were similar in age, body mass index, and LVEF. Prevalence of SDB was higher in males than females. During follow up of 25±10 months, 27% of the population died. Nonsurvivors had lower LVEF (p=0.01), worse NYHA class (p=0.03) a higher proportion of CSR-awake (p<0.001) than survivors.

DETAILED DESCRIPTION:
Bakground: There is little information in sleep disordered breathing (SDB) in women with congestive heart failure (CHF). We studied consecutive CHF patients in order to compare SDB characteristics according to gender, and to determine overall mortality impact of SDB and Cheyne-Stokes respiration (CSR) while awake.

Methods: Eighty nine consecutive outpatients (29 female) with stable CHF (LVEF<45%) were prospectively evaluated. The presence of SDB, as characterized by obstructive sleep apnea (OSA) and CSR during sleep, as well as CSR while awake before sleep onset, were investigated by overnight polysomnography.

ELIGIBILITY:
Inclusion Criteria:

* Patients with resting left ventricular ejection fraction (LVEF) of less than 45% as determined by echocardiography;
* Stable clinical condition as defined by no changes in drug therapy for at least one month before evaluation.

Exclusion Criteria:

* Patients with neurological, pulmonary, renal, musculoskeletal disease, unstable angina, primary valvular heart disease or previous diagnosis of sleep disordered breathing.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Consecutive patients with CHF recruited from the outpatient Heart Failure Unit of the Heart Institute (Instituto do Coraçao do Hospital das Clinicas da Faculdade de Medicina da Universidade de Sao Paulo)
Sampling Method: Non-Probability Sample
Enrollment: 89 (Actual)
Dates: Start 2001-11; Study Completion 2004-03 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Rogerio S Silva, PhD, Principal Investigator — University of Sao Paulo